CLINICAL TRIAL: NCT05127187
Title: Estimation of the Prevalence of HIV, Hepatitis C and Hepatitis B Infection Among Detainees in the Nîmes Administrative Detention Center
Acronym: TRODUMCRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NIMAO/2020-2/MK-1; 2021-A00544-37 (Other: ANSM)
Record Dates: First submitted 2021-11-12; First posted 2021-11-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections; Hepatitis C; Hepatitis B
MeSH Terms: conditions — HIV Infections; Hepatitis C; Hepatitis B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Detainees in an Administrative Detention Center (Experimental)
  Interventions: Diagnostic Test: Rapid diagnosis test against HIV and hepatitis C and B

INTERVENTIONS:
Diagnostic Test: Rapid diagnosis test against HIV and hepatitis C and B — combined Insti VIH® + Toyo VHC®, then First response Ag Hbs tested on capillary blood sample

SUMMARY:
People in Administrative Detention Centers often come from areas of medium or high HIV, hepatitis C & B endemic, and are often unaware of their serological status. Currently, HIV, hepatitis C & B screening is not systematically performed at the CRA of Nîmes, and when performed, serological tests are used. The main disadvantage of this method is the length of time it takes to obtain the results, with subjects frequently discharged before receiving their results.

To improve the care of these vulnerable persons, the aim of this study is to estimate the prevalence of HIV, hepatitis C and hepatitis B in the detainees of the administrative detention center of Nîmes, by systematically screening with a rapid diagnosis test. In case of a positive rapid diagnosis test test, a serology test will confirm the rapid diagnosis test result.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed oral consent
* Patient detained in the Nîmes Administrative Detention Center

Exclusion Criterion

• It is impossible to give the subject informed information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of HIV infection in detainees at the Nîmes Administrative Detention Center | Inclusion
  Rapid diagnosis test: Positive/negative
Prevalence of Hepatitis C infection in detainees at the Nîmes Administrative Detention Center | Inclusion
  Rapid diagnosis test: Positive/negative
Prevalence of Hepatitis B infection in detainees at the Nîmes Administrative Detention Center | Inclusion
  Rapid diagnosis test: Positive/negative

SECONDARY OUTCOMES:
Prevalence of co-infections between HIV, Hepatitis C and Hepatitis B | Inclusion
  Yes or no for co-infection (HIV-Hep C / HIV-Hep B / HepC-HepB / Hiv-HepC-HepB)
Participant country of origin | Inclusion
  Country name
Knowledge of HIV, Hep C and Hep B status | Inclusion
  Yes/no
Participant previous transfusion | Inclusion
  Yes/no
Intravenous drug use | Inclusion
  Yes/no
Intranasal drug use | Inclusion
  Yes/no
Shared drug paraphernalia | Inclusion
  Yes/no
Non-protected sexual activity | Inclusion
  Yes/no
Participant with piercings | Inclusion
  If yes, professional done or not
Participant with tattoos | Inclusion
  If yes, professional done or not
Feasibility of screening | End of study (1 year)
  % of subjects with available samples (ie no subject refusal, subjects arriving at weekend or holiday, study not offered on a weekday, technical problem with test interpretation)
Acceptability of the screening | End of study (1 year)
  % of subjects giving samples

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Kinne, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU Nîmes, Nîmes, France

REFERENCES:
- [Result] Mancy S, Fabbro-Peray P, Alonso S, Berkaoui H, Lambremon L, Vidal H, Hilaire C, Herrmann D, Dapoigny J, Kinne M. Prevalence of HIV, Hepatitis C and Hepatitis B Infection Among Detainees in a French Administrative Detention Centre. J Epidemiol Glob Health. 2024 Sep;14(3):923-932. doi: 10.1007/s44197-024-00238-0. Epub 2024 May 13. PMID 38739355